CLINICAL TRIAL: NCT04304508
Title: Multicenter, Randomized, Placebo-controlled, Double-blind, Parallel Group, Dose-finding Phase 2 Study to Evaluate Efficacy and Safety of BAY2433334 in Patients Following an Acute Non-cardioembolic Ischemic Stroke
Brief Title: Study to Gather Information About Proper Dosing and Safety of the Oral FXIa Inhibitor BAY 2433334 in Patients Following a Recent Non Cardioembolic Ischemic Stroke Which Occurs When a Blood Clot Has Formed Somewhere in the Human Body (But Not in the Heart) Travelled to the Brain.
Acronym: PACIFIC-STROKE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19766; 2019-003431-33 (EudraCT Number)
Record Dates: First submitted 2020-03-08; First posted 2020-03-11 (Actual); Results first posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Acute Non-cardioembolic Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BAY2433334 high dose (Experimental)
  Interventions: Drug: BAY2433334
- BAY2433334 medium dose (Experimental)
  Interventions: Drug: BAY2433334
- BAY2433334 low dose (Experimental)
  Interventions: Drug: BAY2433334
- BAY2433334 matching placebo (Placebo Comparator)
  Interventions: Other: BAY2433334 matching placebo

INTERVENTIONS:
Drug: BAY2433334 — Tablet, taken orally once a day.
  Arms: BAY2433334 high dose; BAY2433334 low dose; BAY2433334 medium dose
Other: BAY2433334 matching placebo — Tablet, taken orally once a day.
  Arms: BAY2433334 matching placebo

SUMMARY:
The purpose of this study is to try to find the best dose of the new drug BAY 2433334 to give to participants and to look at how well BAY 2433334 works on top of antiplatelet therapy in patients following a recent non cardioembolic ischemic stroke which occurs when a blood clot that has not formed in the heart travelled to the brain. BAY 2433334, works by blocking a step of the blood clotting process in our body and thins the blood and is a so called oral FXIa inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 45 years of age and older at the time of signing the informed consent
* Non-cardioembolic ischemic stroke with

  * persistent signs and symptoms of stroke lasting for ≥ 24 hours OR
  * acute brain infarction documented by computed tomography (CT) or MRI AND
  * with the intention to be treated with antiplatelet therapy during the study conduct
* Imaging of brain (CT or MRI) ruling out hemorrhagic stroke or another pathology that could explain symptoms (e.g. brain tumor, abscess, vascular malformation)
* Severity of index event nearest the time of randomization:

  * Part A: minor stroke (defined as National Institutes of Health Stroke Scale (NIHSS) ≤ 7) can be enrolled
  * Part B: participants with minor or moderate stroke and NIHSS ≤ 15 can be enrolled. Participants undergoing thrombolysis or endovascular therapy (mechanical thrombectomy) can be enrolled but at the earliest 24 hours after the intervention
* Randomization within 48 hours after the onset of symptoms of the index event (or after patients were last known to be without symptoms in case of wake-up stroke)
* Ability to conduct an MRI either before randomization or within 72 hours after randomization

Exclusion Criteria:

* Prior ischemic stroke within last 30 days of index event
* History of atrial fibrillation or suspicion of cardioembolic source of stroke
* Dysphagia with inability to safely swallow study medication
* Contraindication to perform brain MRI
* Part A only: thrombolysis or endovascular therapy (mechanical thrombectomy) performed for index event
* Active bleeding; known bleeding disorder, history of major bleeding (intracranial, retroperitoneal, intraocular) or clinically significant gastrointestinal bleeding within last 6 months of randomization.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1808 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (197):
- United States (5):
  - Univ.of South Florida College of Medicine, Tampa, Florida
  - Minneapolis Clinic of Neurology, Ltd., Golden Valley, Minnesota
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - Guilford Neurologic Associates, Greensboro, North Carolina
  - University of Pittsburgh Medical Center Hamot, Erie, Pennsylvania
- Australia (11):
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Grampians Health Ballarat, Ballarat, Victoria
  - Eastern Clinical Research Unit - Box Hill, Box Hill, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - The Alfred Hospital, Prahran, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Austria (7):
  - Krankenhaus der Barmherzigen Brüder Eisenstadt, Eisenstadt, Burgenland
  - Medizinische Universität Innsbruck, Innsbruck, Tyrol
  - Konventhospital Barmherzige Brüder Linz, Linz, Upper Austria
  - Christian-Doppler-Klinik, Salzburg
  - Krankenhaus der Barmherzigen Brüder, Vienna
  - Universitätsklinikum AKH Wien, Vienna
  - Klinik Favoriten - Sozialmedizinisches Zentrum Süd, Vienna
- Belgium (8):
  - Jessa Ziekenhuis, Hasselt, Limburg
  - CHC MontLégia, Liège, Liège
  - AZ Klina / Neurology, Brasschaat
  - UZ Brussel, Brussels
  - UZ Leuven Gasthuisberg, Leuven
  - Kust, Ommeland en Meetjesland (KOM) Network | AZ Damiaan - Neurology Department, Ostend
  - AZ Delta / Neurology, Roeselare
  - Clinique de l'Europe, Uccle
- Bulgaria (10):
  - MHAT Haskovo, Haskovo
  - UMHAT Dr. Georgi Stranski, Pleven
  - MHAT Sveti Pantaleymon - Plovdiv, Plovdiv
  - UMHAT Kanev AD, Rousse
  - First Multiprofile Hospital for Active Treatment Sofia EAD, Sofia
  - MHAT National Cardiology Hospital EAD, Sofia
  - Acibadem City Clinic Multiprofile Hospital for Active Treatm, Sofia
  - UMHATEM N. I. Pirogov EAD, Sofia
  - UMHAT "Sveta Anna"-Sofia, Sofia
  - MHAT Sveta Marina EAD, Varna
- China (8):
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - Baogang hospital, Baotou, Inner Mongolia
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - People's Hospital of Deyang City, Deyang, Sichuan
  - Huashan Hospital, Fudan University, Shanghai
  - Tianjin Huanhu Hospital, Tianjin
- Czechia (9):
  - Fakultni nemocnice u sv. Anny, Brno
  - Nemocnice Ceske Budejovice, a.s. Department of kardiologie, České Budějovice
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Hospital Jihlava - Nemocnice Jihlava, Jihlava
  - Vitkovicka nemocnice a.s., Ostrava Vitkovice
  - Fakultni nemocnice Ostrava, Ostrava-Poruba
  - Nemocnice Pardubickeho kraje, a.s., Pardubicka nemocnice, Pardubice
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Nemocnice na Homolce - Neurology Department, Praha 5-Motol
- Denmark (8):
  - Aalborg Universitetshospital -Neurology, Aalborg
  - Aarhus Universitetshospital, Skejby, Aarhus N
  - Bispebjerg Hospital, Copenhagen
  - Rigshospitalet Glostrup, Glostrup Municipality
  - Herlev Hospital - Neurology Dept., Herlev
  - Regionshospitalet Gødstrup, Herning
  - Nordsjælland Hospital Hillerød, Hillerød
  - Sygehus Lillebaelt | Kolding Sygehus - Medicinske Sygdomme, Kolding
- Finland (3):
  - HUS, Meilahden sairaala, Helsinki
  - Itä-Suomen yliopisto, Kuopio
  - Turun yliopistollinen keskussairaala, Turku
- France (11):
  - Hopital Jean Minjoz, Besançon
  - Hôpital Pellegrin - Bordeaux, Bordeaux
  - Centre Hospitalier Universitaire - Le Kremlin Bicêtre, Le Kremlin-Bicêtre
  - Centre Hospitalier - Le Mans, Le Mans
  - Hôpital B - Lille, Lille
  - Hopital Central - Nancy, Nancy
  - Hôpital Lariboisière - Paris, Paris
  - Hôpital de la Pitié-Salpétrière, Paris
  - Centre hospitalier Sainte Anne, Paris
  - Hôpital Pontchaillou, Rennes
  - Hôpital Purpan - Toulouse, Toulouse
- Germany (11):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Eberhard-Karls-Universität Tübingen, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Rhön-Klinikum Campus Bad Neustadt, Bad Neustadt an der Saale, Bavaria
  - Universitätsklinikum der Johann Wolfgang Goethe Universität, Frankfurt am Main, Hesse
  - Klinikum Frankfurt Höchst GmbH, Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover (MHH), Hanover, Lower Saxony
  - Heinrich-Heine-Universität Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Alfried Krupp Krankenhaus Rüttenscheid /Neurologie, Essen, North Rhine-Westphalia
  - Universitätsklinikum Leipzig AöR, Leipzig, Saxony
  - Klinikum Altenburger Land GmbH, Altenburg, Thuringia
- Hungary (6):
  - Eszak-Pesti Centrumkorhaz-Honvedkorhaz, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Flor Ferenc Korhaz, Kistarcsa
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
  - SZTE ÁOK Szent Györgyi Albert Klinikai Kozpont, Szeged
  - Zala Megyei Szent Rafael Korhaz, Zalaegerszeg
- Italy (9):
  - AUSL di Bologna, Bologna, Emilia-Romagna
  - AUSL della Romagna, Forlì Cesena, Emilia-Romagna
  - AUSL-IRCCS di Reggio Emilia, Reggio Emilia, Emilia-Romagna
  - A.O. San Camillo-Forlanini, Rome, Lazio
  - Ospedale San Raffaele s.r.l., Milan, Lombardy
  - Fondazione Istituto Neurologico Nazionale Casimiro Mondino, Pavia, Lombardy
  - A.O.U. Ospedali Riuniti "Umberto I - G.M.Lancisi - G.Salesi", Ancona, The Marches
  - A.O.U. Senese, Siena, Tuscany
  - A.O. di Perugia, Perugia, Umbria
- Japan (22):
  - Nagoya Ekisaikai Hospital, Nagoya, Aichi-ken
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - St.Mary's Hospital, Kurume, Fukuoka
  - Southern Tohoku Medical Clinic, Kōriyama, Fukushima
  - Hakodate Shintoshi Hospital, Hakodate, Hokkaido
  - Hyogo Prefectural Harima-Himeji General Medical Center, Himeji, Hyōgo
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - JA Toride Medical Center, Toride, Ibaraki
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - Kyoto Okamoto Memorial Hospital, Kusegun, Kyoto
  - Uji-Tokushukai Medical Center, Uji, Kyoto
  - Nozaki Tokushukai Hospital, Daitō, Osaka
  - Kyorin University Hospital, Mitaka, Tokyo
  - Saiseikai Fukuoka General Hospital, Fukuoka
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Gifu Prefectural General Medical Center, Gifu
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Chikamori Hospital, Kochi
  - Saiseikai Kumamoto Hospital, Kumamoto
  - Japanese Red Cross Kumamoto Hospital, Kumamoto
  - Ijinkai Takeda General Hospital, Kyoto
  - Nagano Municipal Hospital, Nagano
- Netherlands (4):
  - Academisch Medisch Centrum (AMC), Amsterdam
  - Zuyderland Medisch Centrum, Heerlen
  - St. Antonius Ziekenhuis, Nieuwegein
  - Isala, Zwolle
- Poland (7):
  - Copernicus PL, M.Kopernik Hospital, Gdansk
  - Samodzielny Publiczny Specjalistyczny Szpital Zachodni, Grodzisk Mazowiecki
  - Gornoslaskie CM im. Prof. Leszka Gieca SUM w Katowicach, Katowice
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Samodzielny Publiczny Szpital Kliniczny nr 4, Lublin
  - Mazowiecki Szpital Specjalistyczny im. dr. Jozefa Psarskiego, Ostrołęka
  - Wojskowy Instytut Medyczny, Warsaw
- Portugal (8):
  - Luz Saude | Hospital Beatriz Angelo - Centro de Investigacao Clinica, Loures, Lisbon District
  - ULSM - Hospital Pedro Hispano, Matosinhos Municipality, Porto District
  - Hospital Garcia de Orta | Research Department, Almada, Setúbal District
  - CHUC - Hospitais da U. Coimbra - Servico de Neurologia, Coimbra
  - CHLO - Hospital Egas Moniz, Lisbon
  - Hospital da Luz - Lisboa, Lisbon
  - CHULN - Hospital Santa Maria, Lisbon
  - CHUSJ - Hospital Sao Joao, Porto
- Russia (8):
  - City Clinical Hospital #3, Chelyabinsk
  - Sci-Res. Institute of Complex Cardiovascular Disorders, Kemerovo
  - Regional Clinical Hospital #1 n.a. prof. S.V. Ochapovsky, Krasnodar
  - Railway clinical hospital on the station Novosibirsk-Glavniy, Novosibirsk
  - City clinical hospital #40 Sestroretsk, Sestroretsk
  - Tomsk Regional Clinical Hospital, Tomsk
  - Clinical Inter-District Hospital of Vsevolozhsk, Vsevolozhsk
  - Sverdlovsk Regional Clinical Hospital #1, Yekaterinburg
- Slovakia (9):
  - Univerzitna nemocnica Bratislava, Nemocnica Stare Mesto, Bratislava
  - Dolnooravska nemocnica s poliklinikou L. Nadasi Jegeho, Dolný Kubín
  - Vseobecna nemocnica s poliklinikou Levoca, a.s., Levoča
  - Liptovska nemocnica s poliklinikou MUDr. Ivana Stodolu, Liptovský Mikuláš
  - Svet zdravia, a. s. Vseobecna nemocnica Rimavska Sobota, Rimavská Sobota
  - Fakultna nemocnica AGEL Skalica, a.s., Skalica
  - Svet zdravia, a.s. Nemocnica s poliklinikou Spisska Nova Ves, Spišská Nová Ves
  - Fakultna nemocnica Trnava, Trnava
  - Vseobecna nemocnica v Ziari nad Hronom, Žiar nad Hronom
- Spain (15):
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela, A Coruña
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de la Mútua de Terrassa, Terrassa, Barcelona
  - Hospital Rey Juan Carlos, Móstoles, Madrid
  - Complejo Hospitalario Universitario de Albacete | Hospital General Universitario - Neurology Department, Stroke Unit, Albacete
  - Hospital del Mar, Barcelona
  - Ciutat Sanitaria i Universitaria de la Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau | Neurology Department - Stroke, No-Cardioembolic-Tia, Barcelona
  - Hospital Universitario Arnau de Vilanova de Lleida, Lleida
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario Ramon y Cajal | Neurology Department - Stroke, No-Cardioembolic-Tia, Madrid
  - Hospital Clinico Universitario San Carlos | Neurologia, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - La Fe University and Polytechnic Hospital | Neurology Service - Vascular Unit, Valencia
  - Hospital Universitario Clinico de Valladolid | Neurology Department, Valladolid
- Sweden (3):
  - Skånes Universitetssjukhus, Lund
  - Danderyds sjukhus, Stockholm
  - Norrlands Universitetssjukhus, Umeå, Umeå
- Switzerland (6):
  - Universitätsspital Basel, Basel, Canton of Basel-City
  - Spitalzentrum Biel, Biel/Bienne, Canton of Bern
  - Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - Kantonsspital Baden, Baden
  - Inselspital Universitätsspital Bern, Bern
  - Ospedale regionale di Lugano, Lugano
- United Kingdom (9):
  - Countess of Chester Hospital, Chester, Cheshire
  - Arrowe Park Hospital, Metropolitan Borough of Wirral, Merseyside
  - Royal Victoria Infirmary, Newcastle upon Tyne, Tyne and Wear
  - Addenbrookes Hospital, Cambridge
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry
  - Glasgow Royal Infirmary | Glasgow Clinical Research Facility, Glasgow
  - Queen Elizabeth University Hospital, Glasgow
  - St George's Hospital, London
  - Charing Cross Hospital, London

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Hart RG, Smith EE, Wang A, Mundl H, Colorado P, Joundi RA, Katsanos AH, Sharma M, Shoamanesh A. Location, size, and risk factors of incident covert brain infarcts in patients with acute non-cardioembolic ischemic stroke: PACIFIC-STROKE trial. Eur Stroke J. 2025 Dec;10(4):1413-1420. doi: 10.1177/23969873251344485. Epub 2025 Jun 13. PMID 40515384
- [Derived] Smith EE, Shoamanesh A, Xu L, Heenan L, Saad F, Colorado P, Chen CH, Lemmens R, De Marchis GM, Caso V, Masjuan J, Hirano T, Milanov I, Campbell BCV, Mas JL, Connolly SJ, Mundl H, Hart RG; PACIFIC-Stroke Steering Committee and Investigators. Effect of the Factor XIa Inhibitor Asundexian According to Baseline Infarct Pattern and on MRI Covert Infarct Outcomes. Stroke. 2024 Feb;55(2):392-402. doi: 10.1161/STROKEAHA.123.043198. Epub 2024 Jan 4. PMID 38174569
- [Derived] Whiteson HZ, Frishman WH. Factor XI/XIa Inhibitors: A New Approach to Anticoagulation. Cardiol Rev. 2025 Jul-Aug 01;33(4):306-311. doi: 10.1097/CRD.0000000000000624. Epub 2023 Dec 1. PMID 38038437
- [Derived] Balali P, Hart RG, Smith EE, Saad F, Colorado P, Lemmens R, De Marchis GM, Caso V, Xu L, Heenan L, Connolly SJ, Mundl H, Shoamanesh A. Cerebral microbleeds and asundexian in non-cardioembolic ischemic stroke: Secondary analyses of the PACIFIC-STROKE randomized trial. Int J Stroke. 2024 Jun;19(5):526-535. doi: 10.1177/17474930231216339. Epub 2023 Dec 16. PMID 37950392
- [Derived] Shoamanesh A, Mundl H, Smith EE, Masjuan J, Milanov I, Hirano T, Agafina A, Campbell B, Caso V, Mas JL, Dong Q, Turcani P, Christensen H, Ferro JM, Veltkamp R, Mikulik R, De Marchis GM, Robinson T, Lemmens R, Stepien A, Greisenegger S, Roine R, Csiba L, Khatri P, Coutinho J, Lindgren AG, Demchuk AM, Colorado P, Kirsch B, Neumann C, Heenan L, Xu L, Connolly SJ, Hart RG; PACIFIC-Stroke Investigators. Factor XIa inhibition with asundexian after acute non-cardioembolic ischaemic stroke (PACIFIC-Stroke): an international, randomised, double-blind, placebo-controlled, phase 2b trial. Lancet. 2022 Sep 24;400(10357):997-1007. doi: 10.1016/S0140-6736(22)01588-4. Epub 2022 Sep 2. PMID 36063821
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 197 centers in 23 countries or regions, between 15-Jun-2020 (first participant first visit) and 18-Feb-2022 (last participant last visit)
Pre-assignment Details: 1880 participants were screened. 72 participants were screening failures. 1808 participants were randomized in a 1:1:1:1 ratio to 4 treatment groups: 455, 450, and 447 participants to asundexian 10 mg, 20 mg and 50 mg groups, 456 participants to placebo group. 22 participants (10, 4, 4 and 4 in the asundexian 10 mg, 20 mg and 50 mg, and placebo groups) never administered.
Groups:
- Asundexian 10 mg: Participants received Asundexian (BAY2433334) 10 mg for 26 weeks at least and up to 52 weeks
- Asundexian 20 mg: Participants received Asundexian (BAY2433334) 20 mg for 26 weeks at least and up to 52 weeks
- Asundexian 50 mg: Participants received Asundexian (BAY2433334) 50 mg for 26 weeks at least and up to 52 weeks
- Placebo: Participants received Asundexian (BAY2433334) placebo for 26 weeks at least and up to 52 weeks
Period: Overall Study
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo
Started (Full analysis set (FAS)) | 455 | 450 | 447 | 456
Treated (Safety analysis set (SAF)) | 445 | 446 | 443 | 452
Completed | 335 (Treatment completed) | 329 (Treatment completed) | 313 (Treatment completed) | 314 (Treatment completed)
Not Completed | 120 | 121 | 134 | 142
Not completed — Subject Decision | 29 | 39 | 37 | 48
Not completed — Death | 6 | 1 | 8 | 5
Not completed — Non-compliance With Study Drug | 3 | 1 | 2 | 0
Not completed — Switching To Other Therapy | 1 | 1 | 1 | 2
Not completed — Subject Decision: COVID-19 Pandemic Related | 0 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 7 | 5 | 11 | 6
Not completed — Logistical Difficulties | 2 | 2 | 3 | 2
Not completed — Missing Information | 1 | 2 | 1 | 3
Not completed — Other | 7 | 6 | 5 | 4
Not completed — Physician Decision: COVID-19 Pandemic Related | 1 | 0 | 0 | 0
Not completed — Physician Decision | 3 | 4 | 9 | 7
Not completed — Study drug never administered | 10 | 4 | 4 | 4
Not completed — Adverse Event | 49 | 50 | 51 | 56
Not completed — Lost to Follow-up | 1 | 5 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS)
Groups:
- Total: Total of all reporting groups
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo | Total
Number analyzed (Participants) | 455 | 450 | 447 | 456 | 1808
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 186 | 154 | 174 | 195 | 709
  >=65 years | 269 | 296 | 273 | 261 | 1099
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 150 | 154 | 150 | 615
  Male | 294 | 300 | 293 | 306 | 1193
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 67 | 67 | 68 | 66 | 268
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 1 | 3
  Black or African American | 4 | 3 | 8 | 3 | 18
  White | 381 | 377 | 367 | 380 | 1505
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 3 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Efficacy-Number of Participants With Composite of Symptomatic Ischemic Stroke or Covert Brain Infarcts Detected by Magnetic Resonance Imaging (MRI)
Description: Ischemic stroke was defined as either of : 1) Rapid onset (or present on awakening) of a new focal neurological deficit with clinical (>24 hours symptoms/signs) or imaging evidence of infarction that was not attributable to a non-ischemic cause; 2) Acute worsening of an existing focal neurological deficit that was judged to be attributable to a new infarction or extension of the previous infarction in the same vascular territory, based on persisting symptoms/signs or imaging evidence of infarction and no evidence of a non-ischemic etiology. If imaging was inconclusive, persistent symptoms/signs must be significant (worsening of NIHSS score of 4 or more) and sustained (duration of ≥24 hours or until death). Covert brain infarcts were defined as incident infarcts detected by serial MRI in the absence of an adjudicated stroke consistent with the location of the infarct. MRI criteria for brain infarction were available in the MRI procedures manual.
Time Frame: From baseline up to 26 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo
Number analyzed (Participants) | 455 | 450 | 447 | 456
Participants
  Symptomatic ischemic stroke | 24 | 25 | 17 | 23
  Covert brain infarct | 56 | 57 | 56 | 55
  Imputed infarcts seen in participants with incomplete MRI follow-up | 6 | 11 | 7 | 5
  Imputed infarcts with the rule of Quan | 11 | 14 | 16 | 15
Statistical Analysis 1: Comparison: Asundexian 10 mg vs Asundexian 20 mg vs Asundexian 50 mg vs Placebo; Dose-response test; Test type: Other — Dose-response test by using multiple comparison procedures (MCP) Mod; p = 0.7976, MCP Mod
Statistical Analysis 2: Comparison: Asundexian 10 mg vs Placebo; Comparison of the Asundexian 10 mg group versus Placebo group; Test type: Other; Crude incidence ratio = 1.044, 90% CI 2-sided [0.8105 to 1.3478]
Statistical Analysis 3: Comparison: Asundexian 20 mg vs Placebo; Comparison of the Asundexian 20 mg group versus Placebo group; Test type: Other; Crude incidence ratio = 1.1963, 90% CI 2-sided [0.9281 to 1.5428]
Statistical Analysis 4: Comparison: Asundexian 50 mg vs Placebo; Comparison of the Asundexian 50 mg group versus Placebo group; Test type: Other; Crude incidence ratio = 1.0485, 90% CI 2-sided [0.8082 to 1.3619]

2. Secondary Outcome: Efficacy-Number of Participants With Composite of Symptomatic Ischemic Stroke and Covert Brain Infarcts Detected by MRI, Cardiovascular (CV) Death, Myocardial Infarction (MI) and Systemic Embolism.
Description: CV death included death due to stroke, MI, heart failure or cardiogenic shock, sudden death or any other death due to other cardiovascular causes. Death due to non-traumatic hemorrhage was included. Acute MI was used when there was evidence of myocardial necrosis in a clinical setting consistent with acute myocardial ischemia. According to MI Universal Definition from 2018 the diagnosis of MI required the combination of: 1) Presence of acute myocardial injury, and 2) Evidence of acute myocardial ischemia derived from the clinical presentation, electrocardiographic changes, or the results of myocardial or coronary artery imaging, or in case of post-mortem pathological findings irrespective of biomarker values. Systemic embolism was defined as abrupt vascular insufficiency associated with clinical or radiological evidence of arterial occlusion in the absence of other likely mechanisms (this did not include thromboembolism of the pulmonary vasculature or venous thrombosis).
Time Frame: From baseline up to 26 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo
Number analyzed (Participants) | 455 | 450 | 447 | 456
Participants
  Ischemic Stroke | 24 | 25 | 17 | 23
  CV death | 3 | 2 | 6 | 6
  MI | 3 | 0 | 3 | 3
  Systemic embolism | 1 | 0 | 0 | 0
  Covert brain infarct | 56 | 57 | 56 | 55
  Imputed infarcts seen in participants with incomplete MRI follow-up | 6 | 11 | 7 | 5

3. Secondary Outcome: Efficacy-Number of Participants With Symptomatic Ischemic Stroke
Description: Definition of symptomatic ischemic stroke can be referred to first Primary endpoint.
Time Frame: From baseline up to 52 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo
Number analyzed (Participants) | 455 | 450 | 447 | 456
Participants | 26 | 26 | 22 | 28

4. Secondary Outcome: Efficacy-Number of Participants With Covert Brain Infarcts Detected by MRI
Description: Definition of covert brain infarcts can be referred to first Primary endpoint.
Time Frame: From baseline up to 26 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo
Number analyzed (Participants) | 455 | 450 | 447 | 456
Participants | 62 | 68 | 63 | 60

5. Secondary Outcome: Efficacy-Number of Participants With Symptomatic Ischemic Stroke, CV Death, MI
Description: Definition of symptomatic ischemic stroke can be referred to first Primary endpoint. Definition of CV death and MI can be referred to first Second endpoint.
Time Frame: From baseline up to 52 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo
Number analyzed (Participants) | 455 | 450 | 447 | 456
Participants | 33 | 30 | 33 | 35

6. Secondary Outcome: Efficacy-Number of Participants With Symptomatic Ischemic and Hemorrhagic Stroke
Description: Definition of symptomatic ischemic can be referred to fourth secondary endpoint. Hemorrhagic stroke was defined as an acute, atraumatic extravasation of blood into the brain parenchyma, intraventricular or subarachnoid space with associated neurological symptoms. This did not include microbleeds or hemorrhagic transformation of an ischemic stroke.
Time Frame: From baseline up to 52 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo
Number analyzed (Participants) | 455 | 450 | 447 | 456
Participants | 26 | 26 | 25 | 30

7. Secondary Outcome: Efficacy-Number of Participants With Disabling Stroke (mRS≥4)
Description: Modified ranking score (mRS): 0-No symptoms at all; 1-No significant disability despite symptoms; despite symptoms, able to carry out all usual duties and activities; 2-Slight disability; unable to carry out all previous activities but able to look after own affairs without assistance; 3-Moderate disability; requiring some help, but able to walk without assistance; 4-Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance; 5-Severe disability; bedridden, incontinent and requiring constant nursing care and attention; 6-Death.
Time Frame: From baseline up to 52 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo
Number analyzed (Participants) | 455 | 450 | 447 | 456
Participants | 5 | 5 | 1 | 3

8. Secondary Outcome: Efficacy-Number of Participants With All-cause Mortality
Time Frame: From baseline up to 52 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo
Number analyzed (Participants) | 455 | 450 | 447 | 456
Participants | 10 | 6 | 17 | 10

9. Primary Outcome: Safety-Number of Participants With Composite of International Society on Thrombosis and Hemostasis (ISTH) Major Bleeding and Clinically Relevant Non-major (CRNM) Bleeding
Description: ISTH Major Bleeding criteria: 1. Fatal bleeding, and/or 2. Symptomatic bleeding in a critical area or organ (intracranial, intraocular, intraspinal, pericardial, retroperitoneal, intraarticular, or intramuscular with compartment syndrome), and/or 3. Clinically overt bleeding associated with a recent decrease in the hemoglobin level of ≥ 2 g/dL (20 g/L; 1.24 mmol/L) compared to the most recent hemoglobin value available before the event, and/or 4. Clinically overt bleeding leading to transfusion of 2 or more units of packed red blood cells or whole blood. ISTH Clinically Relevant Non-Major Bleeding is considered any sign or symptom of hemorrhage that does not fit the criteria for the ISTH definition of major bleeding, but does meet at least one of the following criteria 1. requiring medical intervention by a healthcare professional. 2. leading to hospitalization or increased level of care. 3. prompting a face to face (i.e. not just a telephone or electronic communication) evaluation.
Time Frame: From baseline up to 52 weeks
Population: SAF
Measure: Count of Participants; unit: Participants
Groups:
- Total Asundexian: Asundexian 10 mg group and Asundexian 20 mg group and Asundexian 50 mg
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Total Asundexian | Placebo
Number analyzed (Participants) | 445 | 446 | 443 | 1334 | 452
Participants | 19 | 14 | 19 | 52 | 11
Statistical Analysis 1: Comparison: Asundexian 10 mg vs Placebo; Comparison of the Asundexian 10 mg group versus Placebo group; Test type: Other — Cause specific HRs were only calculated if at least 3 events occurred in 1 of the compared groups and at least 1 event in each of the compared treatment groups; p = 0.1507, Log Rank; Cox Proportional Hazard = 1.724, 90% CI 2-sided [0.924 to 3.215]
Statistical Analysis 2: Comparison: Asundexian 20 mg vs Placebo; Comparison of the Asundexian 20 mg group versus Placebo group; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.5339, Log Rank; Cox Proportional Hazard = 1.285, 90% CI 2-sided [0.662 to 2.494]
Statistical Analysis 3: Comparison: Asundexian 50 mg vs Placebo; Comparison of the Asundexian 50 mg group versus Placebo group; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.1401, Log Rank; Cox Proportional Hazard = 1.749, 90% CI 2-sided [0.938 to 3.262]
Statistical Analysis 4: Comparison: Total Asundexian vs Placebo; Comparison of the Total Asundexian group versus Placebo group; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.1653, Log Rank; Cox Proportional Hazard = 1.585, 90% CI 2-sided [0.918 to 2.736]

10. Secondary Outcome: Safety-Number of Participants With All Bleeding
Description: All bleeding events occurred from first intake of study intervention until 2 days after the last intake of study intervention.
Time Frame: From baseline up to 52 weeks
Population: SAF
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo
Number analyzed (Participants) | 445 | 446 | 443 | 452
Participants | 37 | 48 | 48 | 44

11. Secondary Outcome: Safety-Number of Participants With ISTH Major Bleeding
Description: Definition of ISTH major bleeding can be referred to second Primary endpoint.
Time Frame: From baseline up to 52 weeks
Population: SAF
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo
Number analyzed (Participants) | 445 | 446 | 443 | 452
Participants | 4 | 3 | 7 | 4

12. Secondary Outcome: Safety-Number of Participants With ISTH CRNM Bleeding
Description: Definition of ISTH CRNM bleeding can be referred to second Primary endpoint.
Time Frame: From baseline up to 52 weeks
Population: SAF
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo
Number analyzed (Participants) | 445 | 446 | 443 | 452
Participants | 15 | 12 | 12 | 7

13. Secondary Outcome: Safety-Number of Participants With ISTH Minor Bleeding
Description: All other overt bleeding episodes not meeting the above criteria for ISTH major or CRNM bleeding were classified as minor bleeding (e.g. bleeding from a minor wound that does not prompt a face-to-face evaluation for a physical examination or laboratory testing).
Time Frame: From baseline up to 52 weeks
Population: SAF
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo
Number analyzed (Participants) | 445 | 446 | 443 | 452
Participants | 21 | 39 | 34 | 34

14. Secondary Outcome: Safety-Number of Participants With Intracerebral Hemorrhage (Non-traumatic)
Description: Non-traumatic intracerebral hemorrhage was defined as a hemorrhagic stroke on the "recurrent stroke" CRF page that is in addition classified as a bleeding with bleeding site intracranial (-subarachnoid, -intraparenchymal [excluding microbleeds], or -intraventricular) and spontaneous causality of bleeding, excluding all symptomatic and hemorrhagic transformation (defined by the PT "hemorrhagic transformation").
Time Frame: From baseline up to 52 weeks
Population: SAF
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo
Number analyzed (Participants) | 445 | 446 | 443 | 452
Participants | 0 | 0 | 3 | 1

ADVERSE EVENTS:
Time Frame: After the first administration of study intervention for up to 52 weeks (but not starting after more than 2 days after the last administration). Reporting for the the all-cause mortality considers all deaths that occurred at any time during the study before the last contact, for up to 54 weeks.
Groups:
- Asundexian 10 mg: Subjects received Asundexian (BAY2433334) 10 mg for 26 weeks at least and up to 52 weeks
- Asundexian 20 mg: Subjects received Asundexian (BAY2433334) 20 mg for 26 weeks at least and up to 52 weeks
- Asundexian 50 mg: Subjects received Asundexian (BAY2433334) 50 mg for 26 weeks at least and up to 52 weeks
- Placebo: Subjects received Asundexian (BAY2433334) placebo for 26 weeks at least and up to 52 weeks
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 10/445 | 6/446 | 17/443 | 10/452
Serious Adverse Events (participants affected / at risk) | 90/445 | 83/446 | 93/443 | 98/452
Other Adverse Events (participants affected / at risk) | 126/445 | 127/446 | 136/443 | 136/452
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asundexian 10 mg (N=445) | Asundexian 20 mg (N=446) | Asundexian 50 mg (N=443) | Placebo (N=452)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (3) | 0 (0) | 2 (2) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 4 (4) | 0 (0) | 3 (3)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chordae tendinae rupture (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 3 (3) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Angle closure glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Macular oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal infarction (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intussusception (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomach mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 5 (5) | 4 (4)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angiogram cerebral (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiovascular evaluation (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep study (Investigations) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Liver function test increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Magnetic resonance imaging abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thymoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain stem infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cerebral artery occlusion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 9 (9) | 8 (8) | 9 (10) | 7 (8)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 4 (4) | 0 (0) | 2 (2) | 4 (4)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Haemorrhagic transformation stroke (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Stroke in evolution (Nervous system disorders) | 3 (3) | 4 (4) | 2 (2) | 3 (3)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 9 (9) | 7 (8) | 9 (9) | 13 (14)
Motor dysfunction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Cerebral hypoperfusion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brachial plexopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombotic cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral amyloid angiopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neurological decompensation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cerebral small vessel ischaemic disease (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebellar microhaemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacunar stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemianaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcoholism (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conversion disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial septal defect repair (Surgical and medical procedures) | 5 (5) | 3 (3) | 3 (3) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Carotid endarterectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery bypass (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endarterectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal decompression (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stent placement (Surgical and medical procedures) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Implantable defibrillator insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shoulder arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary angioplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic bypass (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder polypectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder neoplasm surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stent insertion (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Transcatheter aortic valve implantation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vocal cord augmentation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atheroembolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asundexian 10 mg (N=445) | Asundexian 20 mg (N=446) | Asundexian 50 mg (N=443) | Placebo (N=452)
Atrial fibrillation (Cardiac disorders) | 18 (18) | 21 (21) | 16 (16) | 22 (22)
Constipation (Gastrointestinal disorders) | 28 (29) | 18 (20) | 28 (29) | 34 (35)
Diarrhoea (Gastrointestinal disorders) | 12 (12) | 14 (15) | 15 (18) | 12 (12)
Urinary tract infection (Infections and infestations) | 13 (15) | 11 (11) | 13 (14) | 14 (18)
COVID-19 (Infections and infestations) | 22 (22) | 14 (14) | 14 (14) | 12 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (11) | 11 (13) | 16 (16) | 12 (12)
Dizziness (Nervous system disorders) | 7 (7) | 16 (18) | 17 (17) | 14 (14)
Headache (Nervous system disorders) | 19 (20) | 19 (38) | 21 (31) | 18 (19)
Insomnia (Psychiatric disorders) | 6 (6) | 16 (16) | 11 (12) | 12 (13)
Hypertension (Vascular disorders) | 23 (24) | 19 (19) | 25 (25) | 24 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI prohibited from publishing results for 18 months following completion of the study at all sites. Sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review.

DOCUMENTS (2):
  • Study Protocol (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/08/NCT04304508/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/08/NCT04304508/SAP_001.pdf